CLINICAL TRIAL: NCT00811382
Title: Clinical effecT of Heart Failure Management Via Home Monitoring With a Focus on Atrial Fibrillation (effecT)
Acronym: effecT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Criterion according study protocol to end study prematurely was fulfilled.
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS044
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure (HF); Atrial Fibrillation
Keywords: CRT; therapy of AF; telecardiology; home monitoring; cardiovascular hospitalization; cardiovascular mortality
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Masking Description: No Masking.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Access to HMSC (Home Monitoring Service Center) (Experimental): Full functionality of the Home Monitoring System for an early optimization of CRT and management of AF with a full access for the treating physician to the HMSC
  Interventions: Device: Home Monitoring (Cardiac resynchronization therapy and atrial fibrillation therapy, with Home Monitoring feature)
- 2: No access to HMSC (Active Comparator): Limited access of the treating physician to the HMSC where only events regarding implant and lead status will be generated and sent to the physician.
  Interventions: Device: Home Monitoring (Cardiac resynchronization therapy and atrial fibrillation therapy, without Home Monitoring)

INTERVENTIONS:
Device: Home Monitoring (Cardiac resynchronization therapy and atrial fibrillation therapy, with Home Monitoring feature) — Cardiac resynchronization therapy and atrial fibrillation therapy according to medical guidelines, where the physician receives relevant daily data from the implant via Home Monitoring
  Arms: 1: Access to HMSC (Home Monitoring Service Center)
Device: Home Monitoring (Cardiac resynchronization therapy and atrial fibrillation therapy, without Home Monitoring) — Cardiac resynchronization therapy and atrial fibrillation therapy according to medical guidelines, without daily data transmission from the implant via Home Monitoring (except for the safety data on device integrity)
  Arms: 2: No access to HMSC

SUMMARY:
EffecT is a prospective, randomized multicenter study to assess whether management of atrial fibrillation (AF) as well as the early optimization of cardiac resynchronization therapy (CRT) via Home Monitoring decreases mortality and morbidity compared to conventional treatment in subjects with a standard indication for CRT with Implantable Cardioverter Defibrillator (ICD) backup and AF.

DETAILED DESCRIPTION:
EffecT is a prospective, randomized multicenter study to assess whether management of atrial fibrillation as well as the early optimization of cardiac resynchronization therapy via Home Monitoring decreases mortality and morbidity compared to conventional treatment in subjects with a standard indication for CRT with Implantable Cardioverter Defibrillator backup (CRT-ICD) and paroxysmal or persistent AF.

300 patients with a documented history of AF will be enrolled and randomized 1:1 to standard patient management or AF management and early optimization of CRT via Home Monitoring. The patient outcome regarding days lost due to cardiovascular mortality, cardiovascular hospitalization and inappropriate ICD therapy will be documented during an observational period of 1 year.

Another 300 patients undergoing CRT-ICD implantation without a history of AF will undergo an AF evaluation during the first three months of CRT. If a patient shows an AF episode during this period, he is eligible for study inclusion. If no AF episode occurs during AF evaluation, the patient be treated as screening failure.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CRT with ICD-backup
* Paroxysmal or persistent AF
* Optimized HF-related medication

Exclusion Criteria:

* Permanent AF
* Contraindication for anticoagulation
* Stroke within the last 6 weeks
* Acute coronary syndrome within the last 2 months
* Cardiac surgery within the last 2 months
* Acute myocarditis
* Severe chronic obstructive pulmonary disease (COPD)
* Planned cardiac surgery or interventional measures within the coming 3 months
* Dialysis dependency
* Life expectancy < 12 months
* Insufficient GSM (Global System for Mobile Communication)/GPRS (General Packet Radio Service)-network coverage
* Previously implanted unipolar right atrial lead
* Previously implanted right atrial lead with tip-ring distance > 11 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schalij, Prof. Dr., Study Chair — Leiden University Medical Center; Isabelle Van Gelder, Prof. Dr., Study Chair — University of Groningen, The Netherlands; Jan Tijssen, Prof. Dr., Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (21):
- Belgium (2):
  - A.Z. Middelheim, Antwerp
  - AZ St. Jan, Bruges
- Czechia (2):
  - Nemocnice Ceske Budejovice, České Budějovice
  - FN Olomouc, Olomouc
- France (9):
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHRU de Lille, Lille
  - CHRU Hôpital de Villeneuve, Montpellier
  - Hôpital Pasteur, Nice
  - Hôpital La Pitié-Salpetrière, Paris
  - CHU Haut Lévêque, Pessac
  - CHU des Rennes, Hôpital de Pontchaillou, Rennes
  - Hôpital Nord, Saint-Etienne
  - Centre Hospitalier de Rangueil, Toulouse
- Germany (3):
  - Charitè Berlin, Berlin
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - University Hospital, Ulm
- Netherlands (3):
  - Rijnstate Ziekenhuis, Arnhem
  - University Hospital, Groningen
  - University Medical Center, Leiden
- Karolinska University Hospital Stockholm, Stockholm, Sweden
- St. Peter's Hospital, Chertsey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: Access to HMSC: Full functionality of the Home Monitoring System for an early optimization of CRT and management of AF with a full access for the treating physician to the HMSC
  Home Monitoring (CRT and AF therapy with Home Monitoring feature): CRT and AF therapy according to medical guidelines, where the physician receives relevant daily data from the implant via Home Monitoring
- 2: No Access to HMSC: Limited access of the treating physician to the HMSC where only events regarding implant and lead status will be generated and sent to the physician.
  Home Monitoring (CRT and AF therapy, without Home Monitoring): CRT and AF therapy according to medical guidelines, without daily data transmission from the implant via Home Monitoring (except for the safety data on device integrity)
Period: Overall Study
Arm/Group | 1: Access to HMSC | 2: No Access to HMSC
Started | 88 | 75
Completed | 88 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1: Access to HMSC: Full functionality of the Home Monitoring System for an early optimization of CRT and management of AF with a full access for the treating physician to the HMSC.
  Home Monitoring (CRT and AF therapy with Home Monitoring feature): CRT and AF therapy according to medical guidelines, where the physician receives relevant daily data from the implant via Home Monitoring.
- Total: Total of all reporting groups
Arm/Group | 1: Access to HMSC | 2: No Access to HMSC | Total
Number analyzed (Participants) | 88 | 75 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (8.5) | 67.3 (10) | 68.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 67 | 59 | 126
Height,centimeter (cm) [Median (Standard Deviation); unit: cm] | 172 (9) | 171 (8) | 172 (9)
Weight, kilogram (kg) [Mean (Standard Deviation); unit: kg] | 82 (16) | 81 (15) | 81 (15)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (4.4) | 27.6 (4.4) | 27.6 (4.4)
New York Heart Association functional class (NYHA class) [Count of Participants; unit: Participants] — Class I: No limitation of physical activity.
  Class II: Slight limitation of physical activity.
  Class III: Marked limitation of physical activity, but comfortable at rest.
  Class IV: Unable to carry on any physical activity without discomfort and symptoms of heart failure at rest.
  This classification is not an outcome but a patient characteristic at enrollment. From the given explanation, it is obvious that lower classes are better.
  Participants
    Class I | 0 | 0 | 0
    Class II | 7 | 5 | 12
    Class III | 75 | 67 | 142
    Class IV | 6 | 3 | 9
Cardiomyopathy [Number; unit: participants]
  Ischemic | 49 | 40 | 89
  Non-ischemic | 39 | 35 | 74
Left ventricular ejection fraction (LVEF) [Median (Standard Deviation); unit: Percentage %] — The Left ventricular ejection fraction (EF) is always reported in the unit of percentage (%). It is the ratio of pumped blood volume divided by the maximal filling volume. The EF refers to the amount, or percentage, of blood that is pumped (or ejected) out of the ventricles with each contraction.
  An EF of 27 percent means that 27 percent of the total amount of blood in the left ventricle is pushed out with each heartbeat.
  Percentage % | 27 (7) | 26 (7) | 27 (7)
Left Ventricular End-Systolic Volume (LVESV) [Median (Standard Deviation); unit: ml] | 135 (58) | 159 (70) | 146 (64)
Left atrial diameter (LAD) [Mean (Standard Deviation); unit: mm] | 49 (10) | 48 (8) | 48 (9)
Mitral regurgitation [Count of Participants; unit: Participants] — A definition of the severity of Mitral Regurgitation can not be given, because the study did enforce a specific one and physicians used their standard definitions. It is not possible to describe their meaning for laypersons better that with the term used (mild, moderate, severe)
  Participants
    Mild | 38 | 39 | 77
    Moderate | 28 | 15 | 43
    Severe | 3 | 2 | 5
    No regurgitation | 17 | 17 | 34
    not reported | 2 | 2 | 4
History of VT/VF [Number; unit: patients]
  Patients with VT/VF | 22 | 15 | 37
  Patients with No VT/VF | 66 | 60 | 126
QRS duration [Median (Standard Deviation); unit: ms] | 158 (24) | 159 (26) | 158 (25)
Heart Rate [Mean (Standard Deviation); unit: beats/min] | 71 (14) | 68 (16) | 70 (15)
AV (atrioventricular) Block [Number; unit: patients] — The classification of atrioventricular block as 1st, 2nd and 3rd degree follows the standard textbook definition. It is not possible to describe their meaning for laypersons.
  This classification is not outcome but a patient characteristic at enrollment. A lower grade is better.
  patients
    No relevant finding | 36 | 32 | 68
    First Degree | 23 | 17 | 40
    Second Degree | 2 | 3 | 5
    Third Degree | 9 | 4 | 13
    Other | 18 | 19 | 37
Rhythm at enrollment [Number; unit: patients] — Sinus Rhythm: with heart rate in the normal range of 60 - 100 beats/min AF: generally at a rate between 110 and 180 beats/min.
  patients
    Sinus Rhythm | 75 | 66 | 141
    AF | 4 | 6 | 10
    Other | 9 | 3 | 12
Non-CV (cardiovascular) Morbidity at Enrollment [Number; unit: patients] — the sum of participants in all categories for the measure does not equal the overall number of baseline participants due to the fact that patients have sometimes more than 1 non-cv morbidity at enrollment
  patients
    Diabetes mellitus | 35 | 20 | 55
    Renal insufficiency | 15 | 10 | 25
    COPD | 18 | 13 | 31
    Thyroid disease | 15 | 9 | 24
    Hepatic disease | 2 | 1 | 3
    Mental disorder | 4 | 2 | 6
    Other | 28 | 19 | 47
History of AF [Number; unit: patients]
  Paroxysmal | 60 | 47 | 107
  Persistent | 21 | 19 | 40
  no History of AF | 7 | 9 | 16
Ventricular Rate during AF [Mean (Standard Deviation); unit: beats/min] | 104 (33) | 100 (32) | 102 (33)
Days since AF is known [Mean (Standard Deviation); unit: days] | 1222 (2076) | 644 (930) | 974 (1701)
History of pharmacological cardioversion [Number; unit: patients]
  successful | 15 | 9 | 24
  not successful | 5 | 3 | 8
  not tried | 61 | 54 | 115
  not reported | 7 | 9 | 16
History of electrical cardioversion [Number; unit: patients]
  successful | 30 | 24 | 54
  not successful | 1 | 0 | 1
  not tried | 50 | 42 | 92
  not reported | 7 | 9 | 16
History of atrial ablation [Number; unit: patients]
  successful ablation | 0 | 0 | 0
  partly successful | 3 | 3 | 6
  not successful | 3 | 1 | 4
  not tried | 75 | 62 | 137
  not reported | 7 | 9 | 16
History AV node ablation [Number; unit: patients]
  successful | 0 | 1 | 1
  not successful | 1 | 0 | 1
  not tried | 80 | 65 | 145
  not reported | 7 | 9 | 16
AF treatment at enrollment [Number; unit: patients] — some patients underwent both rate control and rhythm control
  patients
    Rate control | 16 | 14 | 30
    Rhythm control | 47 | 37 | 84
    No AF treatment | 21 | 17 | 38
    not reported | 4 | 7 | 11
Medication at Enrollment [Number; unit: patients]
  ACE inhibitor or ARB | 72 | 63 | 135
  Amiodarone | 36 | 36 | 72
  Beta blocker | 69 | 63 | 132
  Calcium channel blocker | 5 | 3 | 8
  Digitalis | 13 | 6 | 19
  Sotalol | 5 | 2 | 7
  Other antiarrhythmic | 1 | 1 | 2
  Anticoagulants | 61 | 54 | 115
  Antiplatelet | 39 | 25 | 64
  Lipid-lowering drug | 63 | 47 | 110
  Nitrate | 7 | 4 | 11
  Spironolactone | 42 | 28 | 70
  Other diuretic | 72 | 63 | 135
  Other medication | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Days Lost
Description: Clinical composite outcome based on the days lost due to cardiovascluar mortality, cardiovascular hospitalization and inappropriate ICD therapy during an observational period of 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Days lost per patient
Arm/Group | 1: Access to HMSC | 2: No Access to HMSC
Number analyzed (Participants) | 88 | 75
Days lost per patient | 15.1 (52.5) | 16.0 (47.8)
Statistical Analysis 1: Comparison: 1: Access to HMSC vs 2: No Access to HMSC; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Heart Failure Clinical Composite Score (Packer Score)
Description: Analysis of the fraction of patients with worsened composite clinical score in the two treatment arms.
Time Frame: 12 months
Population: Endpoint was not evaluated because of the insignificant result for the primary hypothesis and early study discontinuation due to low enrollment
Arm/Group | 1: Access to HMSC (Home Monitoring Service Center) | 2: No Access to HMSC
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Reverse Remodelling (LA Diameter, LVESV, Mitral Regurgitation)
Description: Analysis of the change in left ventricular end-systolic volume, left atrial diameter, left ventricular EF, and the degree of mitral regurgitation from enrollment to the end of the follow-up in the two treatment arms
Time Frame: 12 months
Population: as for outcome 2
Arm/Group | 1: Access to HMSC | 2: No Access to HMSC
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression of AF and AT/AF Burden
Description: The proportion of patients in sinus rhythm or with paroxysmal AF, persistant AF, or permanet AF at the end of the Follow-Up, without statistical evaluation and analysis of AF/AT (atrial tachycardia) burden based on the home monitoring data
Time Frame: 12 months
Population: as for outcome 2
Arm/Group | 1: Access to HMSC | 2: No Access to HMSC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of randomization until the date of death from any cause, study withdrawal, or study termination, which ever came first, assessed up to 1 year
Description: The definition of Adverse Event (AE) and/or serious AE (SAE), used to collect AE information, differs not from the clinicaltrials.gov definitions. There is no source vocabulary for adverse event terms for this study. It is not possible to provide specific AE Terms (e.g. arrhythmia) to indicate whether or not events were related to the device. We used a standard AE Form to document the relationship to the medical device and the investigator ticked "device related, maybe or not related".
Groups:
- 1: Access to HMSC: Full functionality of the Home Monitoring System for an early optimization of cardiac resynchronization therapy and management of atrial fibrillation with a full access for the treating physician to the Home Monitoring Service Center
  Home Monitoring (Cardiac resynchronization therapy and atrial fibrillation therapy with Home Monitoring feature): Cardiac resynchronization therapy and atrial fibrillation therapy according to medical guidelines, where the physician receives relevant daily data from the implant via Home Monitoring
Arm/Group | 1: Access to HMSC | 2: No Access to HMSC
Serious Adverse Events (participants affected / at risk) | 45/88 | 41/75
Other Adverse Events (participants affected / at risk) | 6/88 | 8/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Access to HMSC (N=88) | 2: No Access to HMSC (N=75)
Device related SAEs (Cardiac disorders) | 12 (12) | 9 (11) — It is not possible to provide specific AE Terms to indicate whether or not AEs were related to the device. We used a standard AE Form to document the relationship to the device and the investigator ticked "device related, maybe or not related".
maybe device-related SAEs (Cardiac disorders) | 3 (3) | 0 (0) — It is not possible to provide specific AE Terms to indicate whether or not AEs were related to the device. We used a standard AE Form to document the relationship to the device and the investigator ticked "device related, maybe or not related".
not device-related SAEs (Cardiac disorders) | 39 (73) | 36 (65) — It is not possible to provide specific AE Terms to indicate whether or not AEs were related to the device. We used a standard AE Form to document the relationship to the device and the investigator ticked "device related, maybe or not related".
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Access to HMSC (N=88) | 2: No Access to HMSC (N=75)
device-related AEs (Cardiac disorders) | 5 (19) | 6 (19) — It is not possible to provide specific AE Terms to indicate whether or not AEs were related to the device. We used a standard AE Form to document the relationship to the device and the investigator ticked "device related, maybe or not related".
maybe device-related AEs (Cardiac disorders) | 1 (4) | 2 (4) — It is not possible to provide specific AE Terms to indicate whether or not AEs were related to the device. We used a standard AE Form to document the relationship to the device and the investigator ticked "device related, maybe or not related".

LIMITATIONS AND CAVEATS:
Due to the disappointing enrollment speed, it has been decided to discontinue the study. Therefore, the study is not powered to test the planned hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less